CLINICAL TRIAL: NCT05946005
Title: Effectiveness of Continuous Application of Lidocaine Cream, Povidone Iodine Cream, and Honey on Second-degree Perineal Tear Healing, a Randomized Controlled Clinical Trial
Brief Title: Lidocaine, Povidone Iodine, and Honey Application on Second-degree Perineal Tear Healing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Maisuri Chalid, Head of Maternal Fetal Medicine Division, Department of Obstetrics and Gynecology, Hasanuddin University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UH21110729/2021
Record Dates: First submitted 2023-05-25; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Perineal Tear
Keywords: perineal rupture; lidocaine; povidone-iodine; honey; wound healing; RCT
MeSH Terms: interventions — Honey; Lidocaine; Povidone-Iodine; Control Groups

STUDY DESIGN:
Intervention Model Description: This study was a single-blind randomized control trial conducted at five different hospitals in Makassar from December 2021 to May 2022. All mothers with vaginal delivery who experienced grade II perineal rupture were applied lidocaine cream, povidone iodine cream, honey, and controls, measured on the REEDA and visual analogue scales (VAS) and observed on days 0, 1, 3, 5, 7, and 14. Repeated ANOVA or Friedman tests were used to analyze the data obtained.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Honey (Experimental): Honey is referred to in the Qur'an as a wound healing agent (QS: 16:68 - 69) and has antimicrobial, antioxidant and anti-inflammatory effects. Honey, as an anti-inflammatory, has components of hydrogen peroxide, flavonoids, and phenolic acids that play a role in stimulating angiogenesis (8). Honey also has a high osmolality which provides moisture to the wound, thereby reducing edema and hyperemia and functioning as an antibacterial, so it is expected to reduce the use of antibiotics. Research reported in 2012 stated that honey had the same effect on wound healing and perineal wound pain in postpartum mothers with routine use two times a day for five days (P < 0.05) (9).
  Interventions: Drug: honey
- Lidocaine (Experimental): Lidocaine is used to reduce sensation in the tissues in certain areas. Lidocaine can be injected or applied topically, depending on the need. These topical anesthetics are popular due to their low cost and minimal side effects. The effect of lidocaine on wound healing is still controversial. A study showed the role of lidocaine in wound healing by significantly reducing wound tensile strength on day eight and increasing collagen maturation (7)
  Interventions: Drug: lidocaine
- povidone - iodine (Experimental): Povidone iodine is an antibacterial and anti-inflammatory agent that accelerates wound healing neovascularization. Several studies have used betadine in postpartum mothers with perineal rupture to provide faster wound healing. A study shows that povidone-iodine cream has a better absorption effect on the skin than betadine solution (10).
  Interventions: Drug: povidone-iodine
- control groups (Other): the control group were not given any intervention
  Interventions: Other: control groups

INTERVENTIONS:
Drug: honey — Tresno Joyo honey applied routinely to the wound two times a day for 14 days. BPOM (National Agency of Drug and Food Control) number: MD252109001219
  Other Names: Tresno Joyo honey
  Arms: Honey
Drug: lidocaine — Dolones cream applied routinely to the wound two times a day for 14 days. BPOM (National Agency of Drug and Food Control) number: DKL0922246629AI
  Other Names: Dolones Cream
  Arms: Lidocaine
Drug: povidone-iodine — Betadine cream applied routinely to the wound two times a day for 14 days. BPOM (National Agency of Drug and Food Control) number: PKD20501710037
  Other Names: Betadine cream
  Arms: povidone - iodine
Other: control groups — no intervention is given
  Arms: control groups

SUMMARY:
This clinical trial aims to compare the effectiveness of the continuous application of lidocaine cream, honey, and povidone-iodine cream in second-degree perineal tear healing.

The main question[s] it aims to answer are:

* Which one has better pain relief effectiveness among the three regimens (lidocaine, povidone-iodine, and honey) as measured by the VAS scale
* Which has better wound healing effectiveness among the three regimens as measured by the REEDA scale The study population was postpartum mothers with second-degree perineal rupture who performed vaginal deliveries and sutured perineal ruptures. Each subject will be provided one of the three applications (lidocaine, povidone-iodine, and honey) to be given to their perineal wound.

DETAILED DESCRIPTION:
The sample size was calculated using the formulation for comparative study with power 1 - β = 0.8, two-tail α = 0.05, a mean of the standard deviation of 1.265, and a minimum mean difference of 0.3. The required sample size was 140 sample of labor women (35 samples in each group).

Research subjects included as many as 220 subjects. A total of 215 subjects met the inclusion criteria, consisting of 4 groups based on the type of perineal wound treatment: the group smeared with honey, lidocaine cream, povidone iodine cream, and the control group. There were 5 research subjects who did not meet the criteria, namely: 2 subjects experienced postpartum hemorrhage, 1 subject had a vulvar hematoma and was re-stitched, and 2 subjects were not willing to participate in the study. All study subjects were measured on the REEDA and VAS scales and observed on days 0, 1, 3, 5, 7, and 14. During the observation, 10 subjects could not be followed up further. The research subjects analyzed consisted of honey (n = 50), lidocaine cream (n = 50), povidone-iodine cream (n = 50), and controls (n = 50).

Initially, all participants were assessed for the severity of the wound due to their perineal tear and the VAS pain scale. After that, continuous suturing of the perineum was carried out with Chromic absorbable thread no.2.0 by a competent obstetrician resident according to operational standards. All women with perineal sutures were given ten tablets of paracetamol 500 mg 3 times daily, not antibiotics. After 30 minutes to 1 hour of perineal suturing, the subjects were divided into four groups, each group of at least 50 people was given simple randomized treatment (ratio 1:1:1:1). Each treatment group, i.e. lidocaine cream (Dolones Cream, Sanbe Farma, Indonesia), honey (Madu TJ, Tresno Joyo, Indonesia), povidone-iodine cream (Betadine, Mundi Pharma, Indonesia), and the control group were not given any intervention were applied routinely to the wound two times a day for 14 days and monitored on days 0, 1, 3, 5, 7, and 14. The parameters monitored were the wound healing process and pain scale using the REEDA scale (30 cm ruler) and visual analogue scale (VAS), respectively. The single-blinded method was used to minimize bias. All subjects were given a choice of four closed tubes of different colours, each filled with honey, lidocaine cream and povidone-iodine cream, then given instructions for use by applying twice daily. Monitoring is carried out by providing monitoring cards and being followed daily.

Subjects were taught how to apply it by washing their hands first, then applying it to all perineal wounds. Research subjects were asked to report all complaints and side effects that were felt. All subjects have explained the purpose of the research and confidentiality in data management.

The data were coded, entered, and analyzed using Microsoft Excel 2010 and Statistical Package for the Social Science version 16.0 (SPSS Inc; Chicago, IL, USA). The statistical test used is the ANOVA test if the data is normally distributed or the Kruskal Wallis test if the data is not normally distributed. These two tests were used to compare the three treatment groups. To see the changes in each group, a repeated ANOVA test was used if the data were normally distributed or the Friedman test if the data were not. These tests are used if repeated observations are made more than two times. To find out the normality of the data using the Kolmogorov-Smirnov test. P-value < 0.05 was considered statistically significant. The analyzed data will then be presented as frequency tables, cross-tabulation tables, graphs, and narratives for interpretation and discussion.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in research activities and policy research approval letter.
* Post-partum mothers with second-degree perineal rupture who underwent perineal suturing with episiotomy or spontaneous rupture.

Exclusion Criteria:

* Patients with a history of autoimmunity, cancer, systemic infection, or infection.
* Mother using antibiotics

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation of the Effectiveness of Wound Healing using honey, lidocaine, povidone - iodine and control with the total REEDA ( Redness, Oedema, Ecchymosis, Discharge, Approximation) | 0 - 14 days
  REEDA scale is a tool that assesses the inflammatory process and tissue healing in perineal trauma. Total REEDA scale is calculated and presented, without emphasizing the evaluation of one of the components, namely redness, edema, ecchymosis, discharge, and approximation. Data is presented in numerical scale (0-15). The greater the score is, the less likely the wound appear to heal.
Correlation of the Effectiveness of Wound Healing using honey, lidocaine, povidone - iodine and control with Redness from REEDA scale | 0 - 14 days
  This outcome measures only the redness scale on the REEDA scale. Data is presented in numerical scale (0-3). The greater the score is, the more severe the condition is.
Correlation of the Effectiveness of Wound Healing using honey, lidocaine, povidone - iodine and control with Edema from REEDA scale | 0 - 14 days
  This outcome measures only the edema scale on the REEDA scale. Data is presented in numerical scale (0-3). The greater the score is, the more severe the condition is.
Correlation of the Effectiveness of Wound Healing using honey, lidocaine, povidone - iodine and control with ecchymosis from REEDA scale | 0 - 14 days
  This outcome measures only the ecchymosis scale on the REEDA scale. Data is presented in numerical scale (0-3). The greater the score is, the more severe the condition is.
Correlation of the Effectiveness of Wound Healing using honey, lidocaine, povidone - iodine and control with discharge from REEDA scale | 0 - 14 days
  This outcome measures only the discharge scale on the REEDA scale. Data is presented in numerical scale (0-3). The greater the score is, the more severe the condition is.
Correlation of the Effectiveness of Wound Healing using honey, lidocaine, povidone - iodine and control with approximation from REEDA scale | 0 - 14 days
  This outcome measures only the approximation scale on the REEDA scale. Data is presented in numerical scale (0-3). The greater the score is, the more severe the condition is.

SECONDARY OUTCOMES:
Correlation of the Effectiveness of Reducing Pain Degrees using honey, lidocaine, povidone - iodine and control with the VAS (Visual Analogue Scale) | 0 - 14 days
  VAS is one of the scales that can be used to assess subjective pain presented by an individual. Data is presented in numerical scale (0-10). The greater the score is, the more pain an individual subjectively suffers.
Correlation of the Effectiveness of Decreasing the REEDA Scale and the VAS Scale at the beginning and end of the follow up (all treatment groups: honey, lidocaine, povidone - iodine and control) | 0 - 14 days
  Mean total of REEDA and VAS scales in all treatment group were evaluated and compared at the start and end of follow-up of each individual. Data is presented in numerical scale.

OTHER OUTCOMES:
Age characteristics of study participants | 0 - 14 days
  Age is a measurement of how long individual has lived. In this research, age is classified into several categories. Data is presented in ordinal scale over 3 categories: < 20 years old, 20 - 35 years old, and > 35 years old.
Parity characteristics of study participants | 0 - 14 days
  Parity is a measurement of how many times has an individual given birth. In this research, parity is classified into several categories. Data is presented in categorical scale over 3 categories: primipara (once), multiparous (2-5 times), grand multiparous (> 5 times).
Body mass index characteristics of study participants | 0 - 14 days
  Body mass index is a measurement to assess the nutritional status of an individual. In this research, body mass index is classified into several categories. Data is presented in categorical scale over 2 categories: normal (18.5 - 24.9 kg/m2) and overweight (> 24.9 kg/m2). The classification of the body mass index is accordance with World Health Organization's classification for Asian population.
Blood pressure characteristics of study participants | 0 - 14 days
  Blood pressure is a measurement of the pressure of blood pumped in the human body. In this research, blood pressure is classified into several categories. Data is presented in categorical scale over 2 categories: normotension (systolic BP < 140 mmHg and/or diastolic BP < 90 mmHg) and hypertension (systolic BP >= 140 mmHg and/or diastolic BP >= 90 mmHg)
Anemia characteristics of study participants | 0 - 14 days
  Anemia is a condition where hemoglobin concentration is lower than normal. In this research, anemia is classified into several categories. Data is presented in categorical scale over 3 categories: mild (hemoglobin 10.0 grams/dL to 12.0 grams/dL), moderate (hemoglobin 8.0 - 9.9 grams/dL), and normal (hemoglobin > 12.0 grams/dL).
Episiotomy characteristics of study participants | 0 - 14 days
  Episiotomy is a surgical incision of the perineum and the posterior vaginal wall. In this research, we classify patients whether or not they have undergone the procedure of episiotomy. Data is presented in categorical scale over 2 categories: yes (episiotomy performed) and no (episiotomy not performed).
Birth weight characteristics of study participants | 0 - 14 days
  The weight of the babies delivered. In this research, birth weight is classified into several categories. Data is presented in categorical scale over 2 categories: < 2500 grams, and 2500-4000 grams.
Perineal rupture history characteristics of study participants | 0 - 14 days
  The history whether or not an individual has a history of perineal rupture. Data is presented in categorical scale over 2 categories: yes (a history of perineal rupture was noted) and no (a history of perineal rupture was not noted).

CONTACTS AND LOCATIONS:
Overall Officials: Maisuri Chalid, Phd, Principal Investigator — Hasanuddin University
Locations (1):
- Wahidin Sudirohusodo Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
Because this study has been finished